CLINICAL TRIAL: NCT05161377
Title: Middle Cerebral Artery Aneurysm Trial: A Randomized Care Trial Comparing Surgical and Endovascular Management of MCA Aneurysm Patients
Brief Title: Middle Cerebral Artery Aneurysm Trial
Acronym: MCAAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-00116285
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Middle Cerebral Artery Aneurysm
Keywords: Intracranial aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical management (Active Comparator)
  Interventions: Procedure: Surgical management
- Endovascular management (Active Comparator)
  Interventions: Procedure: Endovascular management

INTERVENTIONS:
Procedure: Surgical management — Surgical clipping will be performed following randomization according to standards of practice, and under general anesthesia. Aneurysms thought by the treating physicians to require deliberate permanent proximal vessel occlusion, construction of a surgical bypass, or other flow-redirecting treatments that do not directly clip the aneurysm will not be excluded; these aneurysms are expected to be more difficult lesions to manage surgically as well as endovascularly.
  Arms: Surgical management
Procedure: Endovascular management — Endovascular treatment will also be performed following randomization, according to standards of practice, and under general anesthesia. Details regarding type of coils, use of adjunctive techniques such as balloon-remodeling, stents, flow-diverters, ISFD/WEBs or other innovative devices, as well as post- treatment medical management issues, will be left up to the physician performing the endovascular treatment and initial strategies determined prior to randomization.
  Arms: Endovascular management

SUMMARY:
Intracranial aneurysms located on the middle cerebral artery (MCA) are considered by many surgeons to represent a distinct subgroup of aneurysms for which clipping may still be the best management option. Most MCA aneurysms are accessible, proximal control can readily be secured in case of rupture, and clip application can typically proceed without requiring the dissection of perforating arteries. In comparison, certain anatomic features of MCA aneurysms such as a wide neck, often including a branch artery origin, frequently render endovascular management more difficult. New endovascular devices were and continue to be introduced to address these anatomic difficulties, including stents, flow diverters, and intra-saccular flow disruptors (ISFDs) such as the WEB. Thus, while most aneurysms are increasingly treated with endovascular methods, many MCA aneurysm patients are still managed surgically, but convincing evidence of which management paradigm is best is lacking.

DETAILED DESCRIPTION:
The subgroup results of ruptured MCA aneurysms taken from ISAT-2 has recently been published. This also suggested that better efficacy could be obtained with surgical management of ruptured MCA aneurysms, with a similar number of residual aneurysms at 1 year in each group (4 surgery, 5 endovascular), but 2 rebleedings from coiled aneurysms (one fatal) and 4 other aneurysms retreated due to growing recurrences discovered on short-term follow-up. Although the ISAT has shown that good-grade, small, anterior circulation aneurysms patients have better 1 year clinical outcomes after being coiled, which was further supported by the Barrow Ruptured Aneurysm Trial (BRAT) study, there are several reasons to suspect that those results do not apply to aneurysms located at the MCA bifurcation. Only 14% of aneurysms in ISAT were on the MCA, likely because lesions in this location were preferentially treated with surgery. Even after selection, the MCA subgroup results were similar for coiling and clipping (RR: 1.01 (0.71-1.45)).

First, the number of selected MCA aneurysm patients included in ISAT was disproportionately small (301/2143 or 14%, as compared to 38% in ISAT-2) and they were recruited between 1994 and 2004, a time when only simple coiling was available. The overall trial result of superior clinical outcomes at 1 year was not confirmed for MCA aneurysms. The clinical primary endpoint of mRS >2 was reached in 39/139 clipped (28.1%, 95% CI:0.21-0.36), and 46/162 coiled patients (28.4%, 95% CI:0.22-0.36).

The suspicion that only selected MCA aneurysm patients were judged eligible for endovascular treatment at the time of ISAT is supported by the pre-randomized BRAT study: Of 61 patients with ruptured MCA aneurysms included between 2003 and 2007, 30 were assigned clipping and 31 coiling. Twenty-one of the 31 (68%) endovascular patients were crossed-over to the surgical arm.15 The Finnish RCT on clipping versus coiling reported only 19 ruptured MCA aneurysms because 59 MCA aneurysm patients were excluded.

If most MCA aneurysms can now be treated endovascularly, clinical results of contemporary technical achievements remain to be properly compared to surgical clipping. In particular, although overall clinical results were similar at one year in ISAT-2, rebleedings and retreatments after endovascular treatment remain worrisome.

The final argument for a new trial dedicated to MCA aneurysms has to do with the eventual interpretation of trial results. ISAT-2 was designed to be, and can still be considered a continuation of the original ISAT trial, with a superiority hypothesis in favor of endovascular treatment. The results presented here suggest that this hypothesis may not be appropriate for ruptured MCA aneurysms. Showing a result for a MCA subgroup that differs from the overall results at the end of ISAT-2 risks being scientifically problematic just as in the original ISAT.

Taken together, the available data and foregoing rationale are sufficient to warrant the conduct of a separate trial of surgical clipping versus endovascular treatment for MCA aneurysms, both ruptured and unruptured. MCAAT will provide a transparent care trial context for clinicians to manage patients with MCA aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* At least one documented, intradural, intracranial aneurysm anywhere on the course of the MCA vessel, ruptured or unruptured. An untreated ruptured aneurysm (with delay in diagnosis) which is suspected to have occurred more than 30 days prior to study inclusion will be considered an unruptured aneurysm
* In the case of SAH, WFNS grade 4 or less
* The patient and aneurysm are considered appropriate for either surgical or endovascular treatment by the treating team

Exclusion Criteria:

* Patients with absolute contraindications administration of contrast material (any type)
* Patients with AVM-associated aneurysms
* Patients or caregivers unable to provide consent
* Poor grade (WFNS 5) ruptured aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Success | up to 5 Years or until death, whichever came first
  The primary composite outcome measure is Treatment Success, a 5-part composite comprising: 1) occlusion or exclusion of the aneurysm using the allocated treatment modality; 2) no intracranial hemorrhage during follow-up; 3) no re-treatment of the target aneurysm during follow-up, 4) no residual aneurysm at 1 year; 5) independence (mRS <3) at 1 year.

SECONDARY OUTCOMES:
The occurrence of an intracranial hemorrhage following treatment | Follow-up for 5 Years or until death, whichever came first
  An intracranial hemorrhage or re-bleed will be judged from cross-sectional imaging (CT or MRI), from a positive lumbar puncture in the setting of an acute headache, or following sudden death preceded by an acute headache.
Failure of aneurysm occlusion using the intended treatment modality | Follow-up for 5 Years or until death, whichever came first
  This will be judged by the treating physician immediately following the attempted treatment.

OTHER OUTCOMES:
Overall mortality | Follow-up for 5 Years or until death, whichever came first
  Mortality from all causes will be recorded, along with cause of death, at one and five years.
Overall morbidity | Follow-up for 5 Years or until death, whichever came first
  Morbidity from all causes will be recorded, at one and five years.
The presence of a residual aneurysm at one year (12 ± 2 months) | at one year (12 ± 2 months)
  This end-point will be determined using non-invasive angiography (CTA or MRA) performed at 12 ± 2 months post-treatment, with all images sent to MCAAT headquarters for Core Lab confirmation.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Darsaut, Principal Investigator — University of Alberta Faculty of Medicine and Dentistry
Locations (1):
- University of Alberta, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Indefinitely

REFERENCES:
- [Derived] Darsaut TE, Keough MB, Boisseau W, Findlay JM, Bojanowski MW, Chaalala C, Iancu D, Weill A, Roy D, Estrade L, Lejeune JP, Januel AC, Carlson AP, Sauvageau E, Al-Jehani H, Orlov K, Aldea S, Piotin M, Gaberel T, Gevry G, Raymond J. Middle Cerebral Artery Aneurysm Trial (MCAAT): A Randomized Care Trial Comparing Surgical and Endovascular Management of MCA Aneurysm Patients. World Neurosurg. 2022 Apr;160:e49-e54. doi: 10.1016/j.wneu.2021.12.083. Epub 2021 Dec 28. PMID 34971833